CLINICAL TRIAL: NCT05442489
Title: Evaluation of the GORE® EXCLUDER® Thoracoabdominal BranchTreatment of the Thoracoabdominal and Pararenal Aortic Aneurysms (TAMBE)
Brief Title: Evaluation of the GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis in the Treatment of the Thoracoabdominal and Pararenal Aortic Aneurysms (TAMBE)
Acronym: TAMBE
Status: Approved for marketing | Type: Expanded Access
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: AAA 17-01 Expanded Access
Record Dates: First submitted 2022-02-21; First posted 2022-07-05 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Thoracoabdominal Aneurysm

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Device: GORE Excluder Thoracoabdominal Branch Endoprosthesis — TEVAR
  Other Names: TAMBE

SUMMARY:
Expanded access tothe GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis is safe and effective in the treatment of thoracoabdominal and pararenal aneurysms.

DETAILED DESCRIPTION:
Gore will permit the use of the TAMBE Device in a manner consistent with the approved CIP provided that its use is needed to treat a serious, but non-life-threatening condition. In the requesting physician's opinion, there must be no acceptable alternative treatment option. Patients are to be consented with an Emergency / Compassionate Use ICF template provided by Gore upon request for this type of device use. Sites will be required to fill out a packet justifying the rationale of use as well as their plan to conduct follow-up surveillance on the non-study subject. Upon performance of the case, the site will immediately notify Gore and provide supporting documentation to facilitate timely, compliant regulatory reporting.

ELIGIBILITY:
• Aortic aneurysm involving the visceral vessels requiring treatment defined as at least one of the following: Fusiform aneurysm diameter ≥ 5 cm Saccular aneurysm (no diameter requirement) Rapid aneurysm growth (≥ 5 mm in one year)

* An Informed Consent Form signed by Subject or legal representative
* Appropriate aortic anatomy to receive the TAMBE Device d

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Keck Medical Center of USC, Los Angeles, California
  - Kaiser Permanente San Francisco Medical Center, San Francisco, California
  - Stanford University, Stanford, California
  - MedStar Health Research Institute - MedStar Washington Hospital, Washington D.C., District of Columbia
  - University of Florida - Gainesville, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan - Cardiac Surgery, Ann Arbor, Michigan
  - Essentia Health, Duluth, Minnesota
  - Division of Vascular Surgery - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Mount Sinai West, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Sanger Heart & Vascular Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPP Heart and Vascular Institute, Pittsburgh, Pennsylvania
  - University of Tennessee -University Vascular Surgeons, Knoxville, Tennessee
  - St. David's Healthcare, Austin, Texas
  - Baylor Heart & Vascular Hospital, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - The Methodist Hospital - Houston, Houston, Texas
  - University of Texas Health Science Center, Houston, Texas
  - Sentara Medical Group, Norfolk, Virginia
  - Carilion Clinic Hospitals, Roanoke, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin
  - Aurora Health Care, Metro Inc., Milwaukee, Wisconsin